CLINICAL TRIAL: NCT07220707
Title: A Pilot Study to Assess the Role of Accelera Stochastic Resonance Wearable Technology to Assist Gait and Mobility in the Older Adult
Brief Title: Wearable Technology to Assist Gait and Mobility in the Older Adult
Status: Not yet recruiting | Type: Observational
Sponsor: Stony Brook University (Other)
Collaborators: Accelera (Unknown)
Responsible Party: Principal Investigator, Randeep Jawa, Professor of Clinical Surgery, Stony Brook University
Other Study IDs: 2025-00142
Record Dates: First submitted 2025-10-20; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Older Adults Who Use an Assistive Device for Mobility
Keywords: older adult; assistive device; stochastic resonance; mobility; gait; fall

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wearing the Accelera device — Wearing the Accelera device prior to retesting gait and mobility

SUMMARY:
This study assesses whether a small wearable ankle bracelet device can improve gait and mobility in the older adult. Before wearing the bracelet, participants will answer a brief questionnaire, have gait and mobility assessed via 3 CDC approved tests and an app, then wear the device and repeat these gait and mobility assessments, and complete a questionnaire.

DETAILED DESCRIPTION:
This is a pilot, observational study with 20 volunteers at Jefferson's Ferry Independent Living. Before the Accelera ankle bracelets are applied, participants will complete a pre-study questionnaire. They will then complete 3 tests that the Centers for Disease Control (CDC) recommends for fall risk assessment, namely the chair stand test, 4-point balance test, and timed up and go test, while using their usual mobility assist devices. If the participants provide optional consent, they will undergo video-based gait/mobility analysis of information derived from the HIPAA compliant Onform video recording app, while they are using their usual mobility assistance devices, if any. In other words, a video recording is made with the app and stored on the apps' HIPAA compliant platform. With the faces obscured, measurements of their gait/mobility will be performed using additional programs as indicated in the Data section. After bracelet application, volunteers will then be encouraged to resume their normal ambulation' (while using their usual mobility assistive devices) for about 30 minutes at the study location as described below. The same 3 tests will be repeated after 30 minutes, along with a post-study questionnaire, and if they consented to video recording above, then repeat videorecording with the Onform video recording app would be performed. With the faces obscured, measurements of their gait/mobility will be performed using additional programs as indicated in the Data section. At this point, the ankle bracelets will be removed - with the subjects having worn them for about 1 hour total. There will be an additional up to 1 hour for completion of the pre- and post-study questionnaires, for a total study session duration of about 1.5 - 2 hours. At each session, we will apply these bracelets to a minimum of 1 patient per session. These sessions will occur at the Wellness Center/gym or other designated area at Jefferson's Ferry 1x per week, with a minimum of one patient for up to 8 patients/week if no holidays, until 20 patients have completed the study. To address infection control, a disposable sock will provide a physical barrier between the device and patient, while still allowing the patient to feel the stochastic resonance.

ELIGIBILITY:
Inclusion Criteria:

1. 65+ years old residing at Independent Living at Jefferson's Ferry
2. Express interest in the ankle wearable device
3. Have capacity as measured by being alert and oriented to person, place, and time
4. Can communicate in English and provide written consent
5. Able to walk and stand unsupported by others and feel ankle vibrations at maximum amplitude.
6. Answers "Yes" to at least one: worry about falling, had a fall within last year, feel unsteady when walking, enrolled in a fall prevention program, or use/have used assistive devices, such as canes or walkers

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Diagnosed with neurodegenerative diseases (such as Parkinson's, Alzheimer's, or Amyotrophic Lateral Sclerosis (ALS))
2. Disability from a stroke or other major neurologic disorder resulting in leg paralysis
3. Active ulcers/rashes/infections on feet or legs, or using orthotics other than arch supports or over the counter knee/ankle supports
4. Significant lymphedema/peripheral edema/or large ankle size that prevents ankle wearable device application or functionality
5. Cannot give written consent
6. Unable to walk today or generally use wheelchairs
7. Unable to participate due to medical or cognitive reasons
8. Any lower extremity amputation other than one toe
9. On anticoagulants or antiplatelet agents other than aspirin
10. Unable to participate due to other medical or cognitive reasons
11. Age under 65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 65+ years who reside at Jefferson's Ferry independent living and generally use assistive devices for mobility, such as a cane or walker.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Performance on mobility/gait assessments and subjective evaluation by participant | from enrollment to the end of the single study session for that participant
  Performance on 3 CDC STEADI tests (timed up and go, chair stand, and 4 point balance test) and mobility as assessed by an optional app and subjective participant assessment on a questionnaire.

SECONDARY OUTCOMES:
sensory thresholds for the device | while wearing the ankle bracelet device
  sensory threshold for the ankle bracelet device

OTHER OUTCOMES:
fall during the study session | during the single study session that the participant is enrolled in
  falls that occur during the study session, while wearing and not wearing the device

CONTACTS AND LOCATIONS:
Locations (1):
- Jefferson's Ferry, South Setauket, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
to protect identity of participants

REFERENCES:
- [Result] Priplata AA, Patritti BL, Niemi JB, Hughes R, Gravelle DC, Lipsitz LA, Veves A, Stein J, Bonato P, Collins JJ. Noise-enhanced balance control in patients with diabetes and patients with stroke. Ann Neurol. 2006 Jan;59(1):4-12. doi: 10.1002/ana.20670. PMID 16287079
- [Result] Priplata AA, Niemi JB, Harry JD, Lipsitz LA, Collins JJ. Vibrating insoles and balance control in elderly people. Lancet. 2003 Oct 4;362(9390):1123-4. doi: 10.1016/S0140-6736(03)14470-4. PMID 14550702
- [Result] Liu W, Lipsitz LA, Montero-Odasso M, Bean J, Kerrigan DC, Collins JJ. Noise-enhanced vibrotactile sensitivity in older adults, patients with stroke, and patients with diabetic neuropathy. Arch Phys Med Rehabil. 2002 Feb;83(2):171-6. doi: 10.1053/apmr.2002.28025. PMID 11833019
- [Result] Galica AM, Kang HG, Priplata AA, D'Andrea SE, Starobinets OV, Sorond FA, Cupples LA, Lipsitz LA. Subsensory vibrations to the feet reduce gait variability in elderly fallers. Gait Posture. 2009 Oct;30(3):383-7. doi: 10.1016/j.gaitpost.2009.07.005. Epub 2009 Jul 25. PMID 19632845
- [Result] Collins JJ, Imhoff TT, Grigg P. Noise-enhanced tactile sensation. Nature. 1996 Oct 31;383(6603):770. doi: 10.1038/383770a0. No abstract available. PMID 8893000

DOCUMENTS (1):
  • Study Protocol: Study Protocol 10-5-25 (2025-10-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT07220707/Prot_000.pdf